CLINICAL TRIAL: NCT03136263
Title: Effects of Oxytocin on Cognitive Control in Adults With Attention Deficit/Hyperactivity Disorder
Brief Title: Oxytocin and Cognitive Control in Adult ADHD
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Elizabeth Austen Lawson, Assistant Professor of Medicine, Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2017P000123
Record Dates: First submitted 2017-04-26; First posted 2017-05-02 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Attention Deficit/Hyperactivity Disorder
Keywords: Attention; Attention deficit/hyperactivity disorder; Cognitive control; Executive control; Executive functions; Impulse control; Impulsivity; Oxytocin
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Impulsive Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Drug order: Oxytocin - placebo (Experimental)
  Interventions: Drug: Oxytocin nasal spray; Drug: Placebo nasal spray
- Drug order: Placebo - oxytocin (Experimental)
  Interventions: Drug: Oxytocin nasal spray; Drug: Placebo nasal spray

INTERVENTIONS:
Drug: Oxytocin nasal spray — Single-dose intranasal oxytocin (24 IU; Syntocinon® nasal spray, Victoria Pharmacy, Zürich, Switzerland)
Drug: Placebo nasal spray — Single-dose intranasal placebo (inactive ingredients of Syntocinon® nasal spray, Victoria Pharmacy, Zürich, Switzerland)

SUMMARY:
This is a randomized, double-blind, placebo-controlled crossover study of single-dose intranasal oxytocin (24 IU) in 18-55 year-old men with attention deficit/hyperactivity disorder (ADHD). Following a screening visit to determine eligibility, participants will return for two main study visits. During the main study visits, study participants will receive either oxytocin (Syntocinon® nasal spray, Victoria Pharmacy, Zürich, Switzerland) or placebo (inactive ingredients of Syntocinon® nasal spray, Victoria Pharmacy), followed by assessments of cognitive control over attention and behavior. Twenty-four participants will be randomized 1:1 to one of two drug orders, i.e., oxytocin - placebo or placebo - oxytocin. In an additional neuroimaging substudy, a subset of participants will undergo task-based and resting-state functional magnetic resonance imaging (fMRI) following oxytocin/placebo administration to investigate the effects of oxytocin on fMRI activation and functional connectivity within the cognitive control network.

ELIGIBILITY:
Inclusion criteria:

* Male
* 18-55 years
* Diagnosis of attention deficit/hyperactivity disorder

Exclusion criteria:

* History of cardiovascular disease (e.g., hypertrophic cardiomyopathy, valvular heart disease, coronary heart disease, or coronary artery spasms)
* History of diabetes mellitus
* Untreated thyroid disease
* Hematocrit below the normal range
* Tobacco use
* Any other significant illness or condition that the investigator determines could interfere with study participation or safety or put the subject at any unnecessary risk
* Excluded at the investigator's clinical judgement of ADHD symptom severity

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2020-11-05 (Actual)

PRIMARY OUTCOMES:
Stop-signal task | First and second main study visits (1-4 weeks apart)
  Mean difference in performance on the stop-signal task between the oxytocin and placebo visits (e.g., stop-signal reaction time)

SECONDARY OUTCOMES:
AX-CPT | First and second main study visits (1-4 weeks apart)
  Mean difference in performance on the AX-CPT between the oxytocin and placebo visits (AY and BX responses)
Category switch task | First and second main study visits (1-4 weeks apart)
  Mean difference in performance on the category switch task between the oxytocin and placebo visits (switch costs and target congruency effect)
Global/local task | First and second main study visits (1-4 weeks apart)
  Mean difference in performance on the global/local task between the oxytocin and placebo visits (global precedence effect)
Simon task | First and second main study visits (1-4 weeks apart)
  Mean difference in performance on the Simon task between the oxytocin and placebo visits (Simon effect and Garner effect)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Lawson, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No